CLINICAL TRIAL: NCT04404088
Title: A Phase II Study of Acalabrutinib, Lenalidomide, and Rituximab (aR2) in Patients With Previously Untreated Follicular Lymphoma
Brief Title: Acalabrutinib, Lenalidomide, and Rituximab for the Treatment of CD20 Positive Stage III-IV, Grade 1-3a Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0034; NCI-2020-01922 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0034 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 3 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 3 Follicular Lymphoma; Grade 3a Follicular Lymphoma
MeSH Terms: interventions — acalabrutinib; Lenalidomide; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, lenalidomide, rituximab) (Experimental): Patients receive acalabrutinib PO BID on days 1-28. Beginning cycle 2, patients receive lenalidomide PO QD on days 1-21 and rituximab IV on days 1, 8, 15, and 22 of cycle 2 and day 1 of subsequent cycles. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Drug: Lenalidomide; Biological: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies how well acalabrutinib, lenalidomide, and rituximab work in treating patients with CD20 positive stage III-IV, grade 1-3a follicular lymphoma. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Giving acalabrutinib, lenalidomide, and rituximab may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of acalabrutinib combined with rituximab and lenalidomide in patients with previously untreated follicular lymphoma (FL) (determined by complete remission [CR] rate by the end of treatment).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of acalabrutinib combined with rituximab and lenalidomide in subjects with FL as assessed by objective response rate (ORR) at the end of treatment, duration of response (DOR), progression rate within 24 months from treatment initiation (progression-free survival [PFS] 24), PFS and overall survival (OS).

II. To evaluate the safety and tolerability of acalabrutinib combined with rituximab and lenalidomide in previously untreated subjects with FL.

EXPLORATORY OBJECTIVE:

I. To determine the pharmacodynamic effects and investigate biomarkers of response and resistance of the 3-drug combination.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Beginning cycle 2, patients receive lenalidomide PO once daily (QD) on days 1-21 and rituximab intravenously (IV) on days 1, 8, 15, and 22 of cycle 2 and day 1 of subsequent cycles. Treatment repeats every 28 days for 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive (+) follicular lymphoma, grade 1, 2, or 3a
* Have had no prior systemic treatment for lymphoma
* Bi-dimensionally measurable disease, with at least one mass lesion >= 2 cm in longest diameter by computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI)
* Meeting Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria for initiation of treatment
* Stage III or IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) >= 1,000/mm^3, independent of growth factor support (within 28 days prior to signing informed consent)
* Platelet counts >= 100,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement with lymphoma, independent of transfusion support in either situation (within 28 days prior to signing informed consent)
* Hemoglobin > 8 g/dL, independent of transfusion support (within 28 days prior to signing informed consent)
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) < 2 x upper limit of normal (ULN) (within 28 days prior to signing informed consent)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula (within 28 days prior to signing informed consent)
* Bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL (within 28 days prior to signing informed consent)
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT) < 1.5 x ULN (within 28 days prior to signing informed consent)
* Must be able to adhere to the study visit schedule and other protocol requirements
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study (females of childbearing potential: must either completely abstain from heterosexual sexual conduct or must use 2 methods of reliable contraception, 1 highly effective [intrauterine device, birth control pills, hormonal patches, injections, vaginal rings, or implants] and at least 1 additional method [condom, diaphragm, cervical cap] of birth control). Reliable contraceptive methods must be started at least 4 weeks before lenalidomide, and continued for at least 4 weeks after last dose of lenalidomide. Males who are sexually active must be practicing complete abstinence or agree to a condom during sexual contact with a pregnant female or female of child bearing potential. Men must agree to not donate sperm during and after the study. For females, these restrictions apply at least 4 weeks before study treatment, during the period of therapy and for 1 month after the last dose of study drug. For males, these restrictions apply during the period of therapy and for 3 months after the last dose of study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study

  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategies (REMS) program
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease, except subjects with a history of central nervous system lymphoma treated and in remission > 6 months
* Evidence of diffuse large B-cell transformation
* Grade 3b FL
* Any prior history of other malignancy besides FL or marginal zone lymphoma, unless the patient has been free of disease for >= 5 years and felt to be at low risk for recurrence by the treating physician, except:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib or lenalidomide capsules, or put the study outcomes at undue risk
* Known history of human immunodeficiency virus (HIV), or active hepatitis C Virus, or active hepatitis B Virus infection, or any uncontrolled active significant infection, including suspected or confirmed John Cunningham (JC) virus infection

  * Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded. Subjects with a history of Hepatitis C who received antiviral treatment are eligible as long as PCR is negative
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Known anaphylaxis or immunoglobulin (Ig) E-mediated hypersensitivity to murine proteins or to any component of acalabrutinib, lenalidomide and/or rituximab
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon). If patients have been on warfarin or equivalent vitamin K antagonists in the past, they will not be eligible if administered within 30 days of the first dose of study drug
* Requires chronic treatment with strong CYP3A inhibitors, for a list of strong CYP3A inhibitors. If patients have been on a strong CYP3A inhibitor in the past, they will not be eligible if the CYP3A inhibitor was administered within 7 days of the first dose of study drug
* Requires chronic treatment with strong CYP3A inducers, for a list of strong CYP3A inducers. If patients have been on a strong CYP3A inducer in the past, they will not be eligible if the CYP3A inducer was administered within 7 days of the first dose of study drug
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association functional classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block
* Active bleeding or known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to study entry
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug
* Patients who have undergone major surgery within 28 days or minor surgery within 3 days of first dose of study drug
* Patients taking corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 10 mg/day prednisone (over these 4 weeks)
* Life expectancy < 6 months
* Neuropathy > grade 1
* Prior exposure to lenalidomide or to a BCR inhibitor, independently from indication
* Patient who require treatment with proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole), and are unable to switch to H2-receptor antagonists
* Patients who have difficulty with or are unable to swallow oral medication, or have disease significantly affecting gastrointestinal function that would limit absorption of oral medication
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Known history of deep vein thrombosis or pulmonary embolism
* Known history of Stevens-Johnson syndrome (SJS) or toxic epidermal necrolysis (TEN) or drug rash with eosinophilia and systemic symptoms (DRESS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | (Up to end of treatment; 1 year)
  Will be based on Cheson, Lugano classification 2014. The number and percentage of subjects with a complete remission at the end of treatment will be tabulated.

SECONDARY OUTCOMES:
Overall response rate (complete response + partial response) | (At the end of treatment ; 1 year )
  Will be based on Cheson, Lugano classification 2014. The number and percentage of subjects with an overall response rate will be tabulated. The best overall response rate will be recorded.
Duration of response | From the time by which measurement criteria for complete response or partial response, whichever is recorded first, is met until death or the first date by which progressive disease is documented, assessed up to 3 years
  Will be based on Cheson, Lugano classification 2014. Cox proportional hazards models will be used to assess the effects of patient prognostic factors on duration of response. Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval.
Progression-free survival within 24 months from treatment initiation | From the treatment start date (cycle 1, day 1) until the firstdate of objectively documented progressive disease or date of death from any cause, assessed up to 24 months
  Will be estimated by the Kaplan-Meier method. Corresponding 95% confidence intervals will be summarized. Cox proportional hazards models will be used to assess the effects of patient prognostic factors on progression-free survival.
Progression-free survival | From the date of cycle 1, day 1 to the date of first documented progression, transformation to diffuse large B-cell lymphoma, initiation of new anti-lymphoma treatment, or death, assessed up to 3 years
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Cox proportional hazards models will be used to assess the effects of patient prognostic factors on progression-free survival.
Overall survival | From the date of cycle 1, day 1 to the date of death regardless of cause, assessed up to 3 years
  Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% confidence interval. Cox proportional hazards models will be used to assess the effects of patient prognostic factors on overall survival.
Frequency, severity, and relatedness of treatment-emergent adverse events (AEs) | Up to 3 years
  Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5. Safety summaries will include tabulations in the form of tables and listings. The frequency (number and percentage) of treatment-emergent AEs will be reported. Additional AE summaries will include AE frequency by AE severity and by relationship to study drug. Clinically significant abnormal laboratory values will be summarized.
Frequency of treatment-emergent AEs requiring study drug discontinuation or dose reduction | Up to 3 years
  Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE version 5. Safety summaries will include tabulations in the form of tables and listings. The frequency (number and percentage) of treatment-emergent AEs will be reported. Additional AE summaries will include AE frequency by AE severity and by relationship to study drug. Clinically significant abnormal laboratory values will be summarized.

OTHER OUTCOMES:
Alteration in immune cell subsets | Up to 3 years
  Will assess whole exome sequencing (WES) of the tissue microenvironment to determine alteration in immune cell subsets. The association between somatic mutations and duration of response will be determined using Cox regression.
Alteration in immune cell subsets | Up to 3 years
  Will assess ribonucleic acid sequencing of tissue microenvironment to determine alteration in immune cell subsets. The frequencies of tumor infiltrating immune cells will be inferred, and their abundance correlated with duration of response.
Cell free circulating deoxyribonucleic acid (DNA) | Up to 3 years
  Will assess cell-free circulating DNA and association with response to therapy. The dynamics of response (i.e. rate of decline of tumor-derived somatic mutations) and ability to achieve negativity of molecular residual disease will be correlated with the duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Strati, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org